CLINICAL TRIAL: NCT00306683
Title: Clinical Assessment of the Treatment With Diazoxide in Children Suffering From Obesity and Hyperinsulinemia Secondary to Surgery of Hypothalamic-pituitary Lesions
Brief Title: Effect of Diazoxide on the Obesity Secondary to Hypothalamic-pituitary Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle BRINDEL, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P040701
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2007-04

CONDITIONS: Hypothalamic-pituitary Lesions; Craniopharyngiomas
Keywords: Hypothalamic-pituitary lesions; Craniopharyngioma; Obesity; Diazoxide; Hyperinsulinemia; Pediatric neurosurgery; Oncology; Pituitary; Hypothalamus
MeSH Terms: conditions — Craniopharyngioma; Obesity; Hyperinsulinism; Neoplasms; Pituitary Diseases | interventions — Diazoxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: DIAZOXIDE

SUMMARY:
In children treated for intracranial lesions, the 2 factors of the obesity are : the location of the lesion (hypothalamic-pituitary region) and craniopharyngiomas

DETAILED DESCRIPTION:
Approximately 80 % of the hypothalamic-pituitary lesions that occur in children are craniopharyngiomas with one or three cases per 1 million children each year.

One major problem remains unsolved : the obesity

This study is performed to optimize the management of the children with hypothalamic-pituitary lesions by reducing the hyperinsulinemia due to the lesion and the surgery

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 18 years
* Obesity with body mass index > 97 percentile or > 2 SD
* Hypothalamic-pituitary lesions not evolutive
* Hyperinsulinemia defined by insulin peak after oral glucose tolerance test>100 UI/L
* Absence of diabetes mellitus defined by basal plasma glucose < 1.2 g/L and glucose peak after oral glucose tolerance test < 2 g/L and HbA1c < 7 %
* Hormonal replacement therapy stable from at least three months excluding the treatment of diabetes insipidus which can be adjusted
* Normal plasma thyroxine
* Written informed consent of the children and the parents

Exclusion Criteria:

* evolutive lesion
* recent surgery or radiotherapy (< 6 months)
* modification of hormonal replacement therapy during the three previous months
* diabetes mellitus defined by basal plasma glucose > 1.2 g/L and glucose peak after oral glucose tolerance test > 2 g/L and HbA1c > 7 %
* renal or hepatic failure
* uncontrolled hypertension
* hypersensitivity to benzothiazine drugs
* pregnancy
* difficulties to understand the protocol

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Relative weight change over two months | 2 months
  Relative weight change over two months
(Weight at Day 1 - Weight at Day 60)/Weight at Day 1

SECONDARY OUTCOMES:
Absolute weight change over two months
Decrease of hyperinsulinemia
Decrease of the glucose peak after oral glucose tolerance test (OGTT)
Evolution of HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Raja BRAUNER, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Kremlin-Bicetre, Paris, France

REFERENCES:
- [Derived] Brauner R, Serreau R, Souberbielle JC, Pouillot M, Grouazel S, Recasens C, Zerah M, Sainte-Rose C, Treluyer JM. Diazoxide in Children With Obesity After Hypothalamic-Pituitary Lesions: A Randomized, Placebo-Controlled Trial. J Clin Endocrinol Metab. 2016 Dec;101(12):4825-4833. doi: 10.1210/jc.2016-2126. Epub 2016 Sep 7. PMID 27603903